CLINICAL TRIAL: NCT01591707
Title: Evaluating a Social and Communication Intervention for Preschoolers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rebecca Landa, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00073501
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorders; school; language; social
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISC+PRT Intervention (Experimental): For the duration of at least one school year children will receive 45-90 minutes of intervention in the classroom in an attempt to increase social and communication skills.
  Interventions: Behavioral: ISC+PRT Intervention
- Instruction As Usual (No Intervention): For the duration of at least one year children will receive the typical classroom instruction

INTERVENTIONS:
Behavioral: ISC+PRT Intervention — Teachers will be trained to implement an intervention in preschool ASD classrooms that provides a learning environment in which social and communication skills are focused on.
  Arms: ISC+PRT Intervention

SUMMARY:
The purpose of this study is to test the effectiveness of a school-based treatment aimed at increasing language and social skills in preschool-aged children with autism spectrum disorder (ASD). Through interactive development (continually seeking educator feedback for intervention improvement) and implementation of the intervention, the investigators hope to provide a feasible and practical means for educators to work with children with ASD in real world, large scale settings. ASD preschool educators, the children enrolled in their classes, between the ages of 3 and 6 years and their families may join.

DETAILED DESCRIPTION:
In Phase 4, KKI staff trained Delaware preschool teachers to serve as model coaches and educators through the Delaware Autism Program. Families whose children were enrolled in participating classrooms were consented through DAP using the school's consent to be videotaped. Any families who did not consent for their child to be videotaped for this training received the nonparticipant consent form currently utilized in this study and staff videotaping took every effort to keep those children out of frame when taping. This cohort involved KKI study team members training 1-2 coaches, who then trained five Delaware school teachers. The IES model was implemented in the teacher's classrooms (n= 5-10 students participating in each classroom; 20-40 children total).

In the current phase of the study, Phase 5 and 6, KKI study team members will continue the evaluation of the IES model, by testing the efficacy of the intervention model in a larger sample (Phase 5) and then analyzing the corresponding data (Phase 6). The larger efficacy study (phase 5) will be conducted on teachers and students recruited from public school districts in Maryland, Delaware, and Pennsylvania using the same IES model and recruitment methods in the previous phases.

ELIGIBILITY:
Inclusion Criteria:

For Teachers:

- Work in an ASD preschool classroom within a cooperating Baltimore County Public School.

For Children:

* Meet Autism Diagnostic Observation Schedule-Generic (ADOS; Lord et al., 2002) and expert clinical judgment criteria for ASD
* Have an IQ or Developmental Quotient of at least 40 based on the Early Learning Composite from the Mullen Scales of Early Learning (Mullen, 1995)
* Be enrolled in a participating Baltimore County Public School ASD preschool classroom
* Be between the ages of 3 and 6 and enrolled in a participating ASD preschool classroom.

Exclusion Criteria:

Children and educators may be taken out of the study if they:

* Are unable to comply with the study protocol
* Change schools due to relocation

Children may also be taken out of this study if they:

* Sustain a head injury or other serious physical injury during the study
* Are not being brought in for testing as designated in the protocol

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2012-07; Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in educator instruction to meet fidelity of intervention. | approximately 4-, 8-, 12-, 16-, 20-, 24-, 28-, 32-, and 36-weeks into the intervention
  Fidelity will be monitored throughout the duration of the intervention by KKI staff to assess the quality and consistency with which educators implement the intervention.

SECONDARY OUTCOMES:
Change in Baseline Autism Diagnostic Observation Schedule | 9 months into treatment
Change in Baseline Mullen Scales of Early Learning | 9 months into treatment
Change in Child's Baseline Spontaneous Imitation Task | 9 months into treatment
Change in Child Classroom-based Social Communication Performance | 9 months into treatment
Change in parent perception of child behavior as recorded by the Autism Composite score of the PDDBI (parent version) | 9 months into treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (3):
- United States (3):
  - Brennen School, Newark, Delaware
  - Kennedy Krieger Institute/Howard County Public Schools, Baltimore, Maryland
  - Elwyn Early Childhood Services, Media, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for teachers will be shared with the Delaware Autism Program to determine feasibility of model implementation. Child participant data will not be shared.